CLINICAL TRIAL: NCT06862635
Title: Efficacy of Hydrotherapy on Balance in Neuropathic Patients Post-Burn
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: MTI University (Other)
Responsible Party: Principal Investigator, Radwa Fayek Hammam, Lecturer at faculty of Physical Therapy, MTI University
Allocation: Not Applicable | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P.T.REC/012/005840
Record Dates: First submitted 2025-02-25; First posted 2025-03-06 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-02

CONDITIONS: Neuropathy; Burn
MeSH Terms: conditions — Burns | interventions — Hydrotherapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Hydrotherapy group (Experimental)
  Interventions: Other: Hydrotherapy
- Land Based exercise group (Active Comparator)
  Interventions: Other: traditional land-based balance exercises

INTERVENTIONS:
Other: Hydrotherapy — Patients will receive hydrotherapy sessions including stretching, resistance, and balance exercises in water
  Arms: Hydrotherapy group
Other: traditional land-based balance exercises — Patients will receive traditional land-based balance exercises in the form of stretching, strengthening and balance exercises.
  Arms: Land Based exercise group

SUMMARY:
Balance problems are common among neuropathic patients following burns, primarily due to sensory and motor impairments.The goal of the study is to investigate the effect of a hydrotherapy program on balance in neuropathic patients following burns. It is a randomized controlled study will be conducted on fifty male patients (age range from 35 to 45 years) with polyneuropathy following lower limb burn injuries, mainly at the sole of the foot, with 3rd-degree injuries and 30% burn extent.

Balance will be assessed before and after treatment using the Biodex Balance System and the Berg Balance Scale (BBS).

Patients will be randomly assigned into two equal groups:

Group A (study group) will receive hydrotherapy sessions including stretching, resistance, and balance exercises in water.

Group B (control group) will receive traditional land-based balance exercises only.

ELIGIBILITY:
Inclusion Criteria:

* polyneuropathy following burn injuries of the lower limb mainly at the sole of the foot.
* 3rd-degree injuries and 30% burn extent.
* Patients' ages range from 35 to 45 years,
* Ability to understand instructions and following commands.

Exclusion Criteria:

* balance disturbances due to neurological disorders other than polyneuropathy (e.g., Parkinson's disease, inner ear disorders, vestibular or cerebellar dysfunctions).
* Uncontrolled hypertension.
* Diabetes mellitus,
* Cognitive impairments
* Blindness.
* Deafness.
* Significant respiratory or cardiac conditions.

Ages: 35 Years to 45 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 50 (Estimated)
Dates: Start 2025-05-05 (Actual); Primary Completion 2025-08-05 (Estimated); Study Completion 2025-08-10 (Estimated)

PRIMARY OUTCOMES:
Balance assessment (Biodex Balance System) | Balance will be assessed by bode balance system before the first session and after 12 sessions (3 months)
  The Biodex Balance System is a multiaxial device that objectively measures and records an individual's ability to stabilize the involved joint under dynamic stress. It uses a circular platform that is free to move in the anterior-posterior and medial-lateral axes simultaneously. It can also be used for the purpose of balance training.

SECONDARY OUTCOMES:
Balance assessment (Berg Balance Scale) | Berg balance scale will be recorded before the fisrt session and after 12 sessions (3 months)
  The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr alainy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No